CLINICAL TRIAL: NCT03756129
Title: A Multi-center, Randomized, subject-and Investigator Blinded, Placebo-controlled, Active Comparator, Parallel-group Proof of Concept Study to Evaluate the Efficacy, Safety, Tolerability and Pharmacokinetics of MIJ821 in Patients With Treatment-resistant Depression
Brief Title: Proof of Concept Study Evaluating the Efficacy and Safety of MIJ821 in Patients With Treatment-resistant Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMIJ821X2201
Record Dates: First submitted 2018-11-13; First posted 2018-11-28 (Actual); Results first posted 2021-05-19 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Depressive Disorder, Treatment-Resistant
Keywords: Refractory Depression; Therapy-Resistant Depression; Treatment Resistant Depression; MDE; MDD; Major depressive disorder (MDD); clinical depression; major depression; unipolar depression; unipolar mood disorder; depression; the blues; mood disorder
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major; Depressive Disorder; Depression; Mood Disorders | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: This is a non-confirmatory, multi-center, 6-treatment arm in the EU countries and 5-treatment arm in the USA (no ketamine arm), randomized, subject and investigator blinded, parallel group, placebo controlled study in treatment-resistant depression patients. The study allows for the inclusion of subjects seeking treatment for their disease from both an 'inpatient' or 'outpatient' clinic setting.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- MIJ821 low dose weekly (Experimental): Infusion. MIJ821 low dose weekly - 0.16 mg/kg
  Interventions: Drug: MIJ821
- MIJ821 low dose bi-weekly (Experimental): Infusion. MIJ821 low dose bi-weekly - 0.16 mg/kg
  Interventions: Drug: MIJ821
- MIJ821 high dose weekly (Experimental): Infusion. MIJ821 high dose weekly - 0.32 mg/kg
  Interventions: Drug: MIJ821
- MIJ821 high dose bi-weekly (Experimental): Infusion. MIJ821 high dose bi-weekly - 0.32 mg/kg
  Interventions: Drug: MIJ821
- Placebo weekly (Placebo Comparator): Infusion. Placebo weekly
  Interventions: Drug: Placebo
- Ketamine 0.5 mg/kg weekly (Active Comparator): Infusion. Ketamine 0.5 mg/kg weekly
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: MIJ821 — Different dosages and different regimen for MIJ821
  Arms: MIJ821 high dose bi-weekly; MIJ821 high dose weekly; MIJ821 low dose bi-weekly; MIJ821 low dose weekly
Drug: Placebo — Infusion
  Arms: Placebo weekly
Drug: Ketamine — Infusion
  Other Names: Ketamine dose to be capped at 40 mg/day for patients over 80 kg
  Arms: Ketamine 0.5 mg/kg weekly

SUMMARY:
This study evaluated the efficacy and safety of the compound MIJ821 compared to placebo in patients aged from 18 to 65 years diagnosed with treatment-resistant depression. The study was conducted in the US and in Europe (Spain). The MIJ821 was administered via infusion on a weekly or bi-weekly basis. The efficacy was measured after 24 hours using a specific golden standard scale, the Montgomery-Asberg Depression Rating Scale. The study duration was 6 weeks of treatment plus 1 month of follow up period.

DETAILED DESCRIPTION:
This was a non-confirmatory, multi-center, 6-treatment arm in European (Spain) and 5-treatment arm in the US (no ketamine arm), randomized, subject and investigator blinded, parallel-group, placebo-controlled study in patients with treatment-resistant depression. The total duration for each subject in the study was maximum 14 weeks: a screening period of maximum 4 weeks, a 36-day treatment period and a 5-week follow-up period.

ELIGIBILITY:
Key Inclusion Criteria:

* Signed informed consent.
* Male and female subjects, 18 to 65 years of age (inclusive) at screening.
* SCID-based DSM-5 defined major depressive episode at the time of screening
* Montgomery-Åsberg Depression Rating Scale (MADRS) score ≥ 24 at screening and baseline
* Failure to respond to two or more antidepressant treatments, where two failed treatments are of two different antidepressants and at least one of which is in the current depressive episode, with adequate dose and duration (≥ 8 weeks duration, doses defined per agent), as identified by the Maudsley Treatment Inventory, and prior psychiatric history, assessed by the investigator, and further documented by medical records and/or third party report (family, friends, clinician-treaters) where available
* If patients are taking any type of psychotropic drugs, a stable dose of psychotropic drugs at screening is defined as no changes in dose or type of antidepressants, antipsychotics, or mood stabilizers for at least 2 weeks prior to screening, if applicable.
* No new antidepressant initiated 4 weeks or less before baseline, and 6 weeks or less before baseline if subject is initiated on fluoxetine
* At least one prior clinical depressive episode (recurrent major depressive disorder), as identified by prior psychiatric history assessed by the investigator, and further documented by medical records and third party report (family, friends, clinician-treaters) where available.
* Able to communicate well, and to understand and comply with study requirements

Key Exclusion Criteria:

* Any current diagnosis of bipolar disorder, schizophrenia, or schizoaffective disorder at screening.
* Current alcohol or substance use disorder (including marijuana and prescribed amphetamine)) meeting DSM-5 criteria, within the past month at baseline. Nicotine and caffeine use disorders will not be considered as exclusionary.
* Prior suicidality caused by or associated with ketamine, as identified by prior psychiatric history assessed by the investigator, and augmented by medical records and third party report (family, friends, clinician-treaters) where available.
* Acute serious and/or imminent suicidal ideation and/or intent within the prior 2 weeks, or any suicide attempt within the prior 4 weeks at screening. Mild to moderate suicidal ideation, using the Sheehan Suicidal Ideation Scale and not meeting the above definition, is not an exclusion criterion.
* Use of other investigational drugs within 30 days or 5 half-lives of randomization, whichever was longer; or longer if required by local regulations at baseline
* Current pregnancy or lactation.
* Positive HIV, Hepatitis B or C test.
* Resting QTcF ≥450 msec (male) or ≥460 msec (female) at pre-treatment baseline
* History of multiple and recurring allergies or allergy to the investigational compound/compound class being used in this study.
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin or in-situ cervical cancer), treated or untreated, within the past 3 years, regardless of whether there is evidence of local recurrence or metastases.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 1 week after stopping of investigational drug.
* History of hypersensitivity to any of the study treatments or excipients or to drugs similar to chemical classes that affect NMDA receptor.
* Current diagnosis of borderline personality disorder or antisocial personality disorder, based on DSM-5 criteria.
* Current acute depressive episode lasting longer than two years continuously, defined as no two week or longer period where depressive symptoms are subsyndromal in severity for a full DSM-5 acute major depressive episode.
* Considered by the investigator, for any other reason, to be an unsuitable candidate for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (8):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Garden Grove, California
  - Novartis Investigative Site, Oakland, California
  - Novartis Investigative Site, Bradenton, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Skokie, Illinois
  - Novartis Investigative Site, Rockville, Maryland
  - Novartis Investigative Site, Berlin, New Jersey
- Spain (4):
  - Novartis Investigative Site, Palma de Mallorca, Balearic Islands
  - Novartis Investigative Site, Vitoria-Gasteiz, Basque Country
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Barcelona

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com/

REFERENCES:
- [Derived] Shelton RC, Litman RE, Hassman H, Walling DP, Ros Montalban S, Salva-Coll J, Zajecka J, Sverdlov O, Gomez-Mancilla B, Healy MP, Shanker YG, Berkheimer M, Faller T, von Raison F, Serban C, Cha JH, Ghaemi SN. Rapid Onset and Sustained Efficacy of Onfasprodil (MIJ821), a Novel NR2B Negative Allosteric Modulator, in Patients With Treatment-Resistant Depression: A Phase 2, Randomized, Placebo-Controlled, Proof-of-Concept Study. J Clin Psychiatry. 2025 Aug 6;86(3):23m15246. doi: 10.4088/JCP.23m15246. PMID 40767837
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=721

RESULTS

PARTICIPANT FLOW:
Groups:
- MIJ821 0.16 mg/kg Weekly: MIJ821 0.16 mg/kg weekly
- MIJ821 0.16 mg/kg Biweekly: MIJ821 0.16 mg/kg biweekly
- MIJ821 0.32 mg/kg Weekly: MIJ821 0.32 mg/kg weekly
- MIJ821 0.32 mg/kg Biweekly: MIJ821 0.32 mg/kg biweekly
- Ketamine 0.5 mg/kg Weekly: Ketamine 0.5 mg/kg weekly
- Placebo Weekly: Placebo weekly
Period: Overall Study
Arm/Group | MIJ821 0.16 mg/kg Weekly | MIJ821 0.16 mg/kg Biweekly | MIJ821 0.32 mg/kg Weekly | MIJ821 0.32 mg/kg Biweekly | Ketamine 0.5 mg/kg Weekly | Placebo Weekly
Started | 11 | 10 | 10 | 9 (1 participant in this group was randomized but not treated, and is not included in this data set.) | 10 (1 participant in this group was randomized but not treated, and is not included in this data set.) | 20
Completed | 8 | 8 | 7 | 6 | 9 | 15
Not Completed | 3 | 2 | 3 | 3 | 1 | 5
Not completed — Adverse Event | 1 | 1 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 3 | 1 | 1 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MIJ821 0.16 mg/kg Weekly | MIJ821 0.16 mg/kg Biweekly | MIJ821 0.32 mg/kg Weekly | MIJ821 0.32 mg/kg Biweekly | Ketamine 0.5 mg/kg Weekly | Placebo Weekly | Total
Number analyzed (Participants) | 11 | 10 | 10 | 9 | 10 | 20 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 9 | 10 | 9 | 10 | 20 | 69
  >=65 years | 0 | 1 | 0 | 0 | 0 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.6 (11.70) | 53.7 (9.33) | 42.9 (14.47) | 46.6 (11.83) | 52.3 (6.96) | 44.8 (10.69) | 47.7 (11.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 6 | 6 | 7 | 9 | 35
  Male | 9 | 5 | 4 | 3 | 3 | 11 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 4 | 4 | 8 | 0 | 10 | 29
  White | 8 | 6 | 6 | 1 | 9 | 9 | 39
  More than one race | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Total Score of the Montgomery Asberg Depression Rating Scale (MADRS) at 24 Hrs
Description: Efficacy. To assess change from baseline in the total MADRS score. The efficacy of MIJ821 in treatment-resistant depression will be compared to the placebo after single dose administration. MADRS is a clinician-rated scale designed to measure depression severity and detects changes due to antidepressant treatment: the test consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition.
Time Frame: Baseline, and at 24 hours
Population: Intent to Treat analysis set
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Groups:
- Pooled MIJ821 0.16 mg/kg: Pooled MIJ821 0.16 mg/kg
- Pooled MIJ821 0.32 mg/kg: Pooled MIJ821 0.32 mg/kg
Arm/Group | Pooled MIJ821 0.16 mg/kg | Pooled MIJ821 0.32 mg/kg | Ketamine 0.5 mg/kg Weekly | Placebo Weekly
Number analyzed (Participants) | 21 | 19 | 10 | 20
Scores on a Scale | -15.51 (1.9) | -12.98 (1.9) | -12.94 (2.7) | -7.27 (1.9)
Statistical Analysis 1: Comparison: Pooled MIJ821 0.16 mg/kg vs Placebo Weekly; Comparison of adjusted arithmetic mean: Mean Difference: "Pooled MIJ821 0.16 mg/kg" minus "placebo". The MIJ821 treatment arms vs placebo are primary; Test type: Superiority; p = 0.0013, ANCOVA; Median Difference (Net) = -8.25, 80% CI 2-sided [-11.67 to -4.83]
Statistical Analysis 2: Comparison: Pooled MIJ821 0.32 mg/kg vs Placebo Weekly; Comparison of adjusted arithmetic mean: Mean Difference: "Pooled MIJ821 0.32 mg/kg" minus "placebo". The MIJ821 treatment arms vs placebo are primary; Test type: Superiority; p = 0.0196, ANCOVA; Mean Difference (Net) = -5.71, 80% CI 2-sided [-9.22 to -2.20]

2. Secondary Outcome: Change From Baseline in the Total Score of the Montgomery Asberg Depression Rating Scale (MADRS) at 48 Hrs
Description: as for outcome 1
Time Frame: Baseline, and at 48 hours
Population: Intent to Treat analysis set. Please note that some participants missed some visits in the study, and thus data for this outcome measure were not collected for some participants.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Pooled MIJ821 0.16 mg/kg | Pooled MIJ821 0.32 mg/kg | Ketamine 0.5 mg/kg Weekly | Placebo Weekly
Number analyzed (Participants) | 19 | 16 | 4 | 19
Scores on a Scale | -14.94 (2.2) | -15.25 (2.4) | -18.89 (4.8) | -7.88 (2.2)
Statistical Analysis 1: Comparison: Pooled MIJ821 0.16 mg/kg vs Placebo Weekly; Comparison of adjusted arithmetic mean: Mean Difference: "Pooled MIJ821 0.16 mg/kg" minus "placebo"; Test type: Superiority; p = 0.0130, ANCOVA; Mean Difference (Net) = -7.06, 80% CI 2-sided [-11.06 to -3.06]
Statistical Analysis 2: Comparison: Pooled MIJ821 0.32 mg/kg vs Placebo Weekly; Comparison of adjusted arithmetic mean: Mean Difference: "Pooled MIJ821 0.32 mg/kg" minus "placebo"; Test type: Superiority; p = 0.0133, ANCOVA; Median Difference (Net) = -7.37, 80% CI 2-sided [-11.57 to -3.18]

3. Secondary Outcome: Change From Baseline in the Total Score of the Montgomery Asberg Depression Rating Scale (MADRS) at Week 6
Description: as for outcome 1
Time Frame: Baseline, and at Week 6
Population: Intent to Treat analysis set
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | MIJ821 0.16 mg/kg Weekly | MIJ821 0.16 mg/kg Biweekly | MIJ821 0.32 mg/kg Weekly | MIJ821 0.32 mg/kg Biweekly | Ketamine 0.5 mg/kg Weekly | Placebo Weekly
Number analyzed (Participants) | 8 | 8 | 8 | 6 | 9 | 17
Scores on a Scale | -12.71 (3.4) | -14.08 (3.4) | -13.04 (3.5) | -10.68 (3.9) | -12.86 (3.3) | -7.62 (2.3)
Statistical Analysis 1: Comparison: MIJ821 0.16 mg/kg Weekly vs Placebo Weekly; Comparison of adjusted arithmetic mean: Mean Difference: "MIJ821 0.16 mg/kg weekly" minus "placebo"; Test type: Superiority; p = 0.1082, ANCOVA; Mean Difference (Net) = -5.09, 80% CI 2-sided [-10.37 to 0.19]
Statistical Analysis 2: Comparison: MIJ821 0.32 mg/kg Weekly vs Placebo Weekly; Comparison of adjusted arithmetic mean: Mean Difference: "MIJ821 0.32 mg/kg weekly" minus "placebo"; Test type: Superiority; p = 0.0993, ANCOVA; Mean Difference (Net) = -5.42, 80% CI 2-sided [-10.83 to -0.02]
Statistical Analysis 3: Comparison: MIJ821 0.16 mg/kg Biweekly vs Placebo Weekly; Comparison of adjusted arithmetic mean: Mean Difference: "MIJ821 0.16 mg/kg biweekly" minus "placebo"; Test type: Superiority; p = 0.0598, ANCOVA; Mean Difference (Net) = -6.46, 80% CI 2-sided [-11.78 to -1.15]
Statistical Analysis 4: Comparison: MIJ821 0.32 mg/kg Biweekly vs Placebo Weekly; Comparison of adjusted arithmetic mean: Mean Difference: "MIJ821 0.32 mg/kg biweekly" minus "placebo"; Test type: Superiority; p = 0.2491, ANCOVA; Mean Difference (Net) = -3.06, 80% CI 2-sided [-8.86 to 2.74]

4. Secondary Outcome: Change From Baseline in the Young Mania Rating Scale
Description: To assess risk of mania induction. The Young Mania Rating Scale has 11 items and is based on the patient's subjective report of his/her clinical condition over the previous 48 hours. There are 4 items that are scored from 0 to 8 (irritability, speech, thought content, and disruptive/aggressive behavior) and the remaining items are scored from 0 to 4. Higher scores indicate more severe mania.
  The total clinical score was calculated as the summation of the individual subscale scores. The maximum for the total YMRS score is 60. The range is 0 to 60 with the higher score indicating more severe symptoms.
Time Frame: Baseline, 24 hours, and 6 weeks (day 43)
Population: Intent-to-treat analysis set. The number of participants analyzed varies from one visit to another because of missed visits and early terminations.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | MIJ821 0.16 mg/kg Weekly | MIJ821 0.16 mg/kg Biweekly | MIJ821 0.32 mg/kg Weekly | MIJ821 0.32 mg/kg Biweekly | Ketamine 0.5 mg/kg Weekly | Placebo Weekly
Number analyzed (Participants) | 11 | 10 | 10 | 9 | 10 | 20
Scores on a Scale
  Adjusted arithmetic mean change from baseline at 24 hrs (n=11,10,10,9,10,20) | -1.41 (0.5) | -1.07 (0.5) | -1.66 (0.5) | -0.81 (0.5) | -1.56 (0.5) | -0.72 (0.3)
  Adjusted arithmetic mean change from baseline at day 43 (n=8,8,8,6,9,17): number analyzed (Participants) | 8 | 8 | 8 | 6 | 9 | 17
  Adjusted arithmetic mean change from baseline at day 43 (n=8,8,8,6,9,17) | -1.28 (0.6) | -2.13 (0.7) | -0.65 (0.7) | -1.55 (0.7) | -1.80 (0.7) | -0.92 (0.4)

5. Secondary Outcome: Bech-Rafaelsen Melancholia Scale
Description: To assess efficacy in the melancholic subtype of depression. Depression scales are used primarily to measure changes, for example, to evaluate the efficacy of treatment with antidepressants. The Bech-Rafaelsen Melancholia Scale (BRMS) is a frequently used clinician rating scale to assess the severity of depression over the past 3 days. Each of the 11 BRMS items is operationally defined on a five-point scale (0-4); hence, the total score ranges from 0 to 44, higher scores indicating greater severity of depression.
Time Frame: Baseline, 24 hours, 48 hours and 6 weeks (Day 43)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | MIJ821 0.16 mg/kg Weekly | MIJ821 0.16 mg/kg Biweekly | MIJ821 0.32 mg/kg Weekly | MIJ821 0.32 mg/kg Biweekly | Ketamine 0.5 mg/kg Weekly | Placebo Weekly
Number analyzed (Participants) | 11 | 10 | 10 | 9 | 10 | 20
Scores on a Scale
  Change at 24 hrs (n=11,10,10,8,9,20): number analyzed (Participants) | 11 | 10 | 10 | 8 | 9 | 20
  Change at 24 hrs (n=11,10,10,8,9,20) | -11.9 (5.941) | -9.5 (4.625) | -7.9 (6.903) | -8.1 (4.612) | -7.7 (5.766) | -6.0 (5.262)
  Change at 48 hrs (n=9,10,9,7,4,19): number analyzed (Participants) | 9 | 10 | 9 | 7 | 4 | 19
  Change at 48 hrs (n=9,10,9,7,4,19) | -9.9 (5.326) | -8.0 (5.185) | -7.6 (8.383) | -8.0 (5.508) | -12.5 (7.853) | -6.7 (6.659)
  Change at day 43 (n=8,8,8,6,9,17): number analyzed (Participants) | 8 | 8 | 8 | 6 | 9 | 17
  Change at day 43 (n=8,8,8,6,9,17) | -8.6 (6.589) | -8.6 (5.423) | -7.6 (10.013) | -6.0 (9.338) | -8.9 (8.343) | -6.9 (5.988)

6. Secondary Outcome: PK Properties of MIJ821 in Plasma - Cmax (ng/mL)
Description: To assess MIJ821 pharmacokinetics in plasma described by Cmax. A single, sparse PK measurement was taken on Day 1.
Time Frame: Day 1
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Pooled MIJ821 0.16 mg/kg | Pooled MIJ821 0.32 mg/kg
Number analyzed (Participants) | 14 | 11
ng/mL | 99.5 (47.8) | 149 (63.4)

7. Secondary Outcome: PK Properties of MIJ821 in Plasma - Tmax (ng/mL)
Description: To assess MIJ821 pharmacokinetics in plasma described by Tmax. A single, sparse PK measurement was taken on Day 1.
Time Frame: Day 1
Population: PK analysis set
Measure: Median (Full Range); unit: hour
Arm/Group | Pooled MIJ821 0.16 mg/kg | Pooled MIJ821 0.32 mg/kg
Number analyzed (Participants) | 14 | 11
hour | 0.683 [0.650 to 0.700] | 0.667 [0.667 to 0.700]

8. Secondary Outcome: PK Properties of MIJ821 in Plasma - AUClast (h*ng/mL)
Description: To assess MIJ821 pharmacokinetics in plasma described by AUClast (h*ng/mL). A single, sparse PK measurement was taken on Day 1.
Time Frame: Day 1
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Pooled MIJ821 0.16 mg/kg | Pooled MIJ821 0.32 mg/kg
Number analyzed (Participants) | 14 | 11
h*ng/mL | 496 (239) | 738 (302)

9. Secondary Outcome: PK Properties of MIJ821 in Plasma - AUC0-24h (h*ng/mL)
Description: To assess MIJ821 pharmacokinetics in plasma described by AUC0-24h (h*ng/mL). A single, sparse PK measurement was taken on Day 1.
Time Frame: Day 1
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Pooled MIJ821 0.16 mg/kg | Pooled MIJ821 0.32 mg/kg
Number analyzed (Participants) | 13 | 11
h*ng/mL | 462 (232) | 713 (275)

10. Secondary Outcome: Change From Baseline in the CORE Melancholia Total Scale
Description: To assess efficacy in melancholic subtype of depression. This scale is an 18 item scale, with a 6 item component capturing cognitive impairment and two motoric scales capturing psychomotor retardation (7 items) and psychomotor agitation (5 items). A cut-off score of 8 or more has been shown to ifferentiate melancholic from non-melancholic depression, with higher scores representing a greater probability of melancholic depression. (Parker and McCraw 2017).
  The total clinical score was calculated as the summation of the individual subscale scores. The maximum for the total CORE Melancholia score is 54. The range is 0 to 54 with the higher score indicating more severe symptoms.
Time Frame: Baseline, 24 hours, 48 hrs, and 6 weeks (day 43)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | MIJ821 0.16 mg/kg Weekly | MIJ821 0.16 mg/kg Biweekly | MIJ821 0.32 mg/kg Weekly | MIJ821 0.32 mg/kg Biweekly | Ketamine 0.5 mg/kg Weekly | Placebo Weekly
Number analyzed (Participants) | 11 | 10 | 10 | 9 | 10 | 20
Scores on a Scale
  Adjusted arithmetic mean change from baseline at 24 hrs (n=4,3,4,3,9,8): number analyzed (Participants) | 4 | 3 | 4 | 3 | 9 | 8
  Adjusted arithmetic mean change from baseline at 24 hrs (n=4,3,4,3,9,8) | -4.76 (2.9) | -3.64 (3.6) | -3.93 (3.0) | 1.38 (3.5) | -5.07 (2.0) | -3.61 (2.0)
  Adjusted arithmetic mean change from baseline at 48 hrs (n=2,3,3,2,4,9): number analyzed (Participants) | 2 | 3 | 3 | 2 | 4 | 9
  Adjusted arithmetic mean change from baseline at 48 hrs (n=2,3,3,2,4,9) | -5.77 (3.9) | -2.82 (3.7) | -5.92 (3.2) | 1.62 (4.0) | -6.68 (2.6) | -5.06 (1.9)
  Adjusted arithmetic mean change from baseline at day 43 (n=3,2,3,2,8,8): number analyzed (Participants) | 3 | 2 | 3 | 2 | 8 | 8
  Adjusted arithmetic mean change from baseline at day 43 (n=3,2,3,2,8,8) | -5.79 (3.4) | -4.82 (4.4) | -7.24 (3.5) | -6.49 (4.3) | -9.01 (2.1) | -5.21 (2.1)

11. Secondary Outcome: Summary of Adverse Events
Description: Summary of Adverse Events
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 30 post treatment, up to a maximum duration of 66 days.
Population: safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | MIJ821 0.16 mg/kg Weekly | MIJ821 0.16 mg/kg Biweekly | MIJ821 0.32 mg/kg Weekly | MIJ821 0.32 mg/kg Biweekly | Ketamine 0.5 mg/kg Weekly | Placebo Weekly
Number analyzed (Participants) | 11 | 10 | 10 | 9 | 10 | 20
Participants
  AEs, subjects with AEs | 7 | 6 | 7 | 6 | 6 | 7
  Study drug-related AEs | 5 | 5 | 7 | 5 | 6 | 5
  SAEs | 0 | 1 | 0 | 3 | 0 | 1
  AEs leading to discontinuation of study treatment | 1 | 0 | 0 | 2 | 0 | 1
  Study drug-related AEs leading to discontinuation of study treatment | 0 | 0 | 0 | 0 | 0 | 1

12. Secondary Outcome: Clinician-Administered Dissociative States Scale
Description: To assess safety and tolerability, especially dissociative side effects. The Clinical-Administered Dissociative States Scale (CADSS) is a questionnaire that assesses dissociative effects. Each item is scored from 0 to 4 and individual scores are to be summed to obtain a total score ranging from a minimum of 0 to a maximum of 80. Higher scores represent a more severe condition.
Time Frame: Change from baseline at 24 hours, 48 hours, and 6 weeks (Day 43)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | MIJ821 0.16 mg/kg Weekly | MIJ821 0.16 mg/kg Biweekly | MIJ821 0.32 mg/kg Weekly | MIJ821 0.32 mg/kg Biweekly | Ketamine 0.5 mg/kg Weekly | Placebo Weekly
Number analyzed (Participants) | 11 | 10 | 10 | 9 | 10 | 20
Scores on a Scale
  Change at 24 hrs (n=11,10,10,8,10,20): number analyzed (Participants) | 11 | 10 | 10 | 8 | 10 | 20
  Change at 24 hrs (n=11,10,10,8,10,20) | 1.09 (5.262) | 1.10 (2.726) | 2.10 (3.414) | 3.00 (3.703) | -0.50 (0.707) | -0.25 (0.716)
  Change at 48 hrs (n=9,10,9,7,4,19): number analyzed (Participants) | 9 | 10 | 9 | 7 | 4 | 19
  Change at 48 hrs (n=9,10,9,7,4,19) | -0.22 (0.667) | 0.50 (2.369) | 4.44 (10.394) | 3.14 (3.976) | 0.00 (0.00) | -0.16 (0.375)
  Change at day 43 (n=8,8,8,6,9,17): number analyzed (Participants) | 8 | 8 | 8 | 6 | 9 | 17
  Change at day 43 (n=8,8,8,6,9,17) | 0.00 (1.927) | 0.00 (0.00) | 0.38 (1.061) | 1.00 (2.449) | 0.00 (1.118) | -0.18 (0.636)

13. Secondary Outcome: Change From Baseline in the Dissociative Experiences Total Score
Description: The Dissociative Experiences Scale (DES) consists of twenty-eight questions about experiences the subject has experienced in his/her daily life. The subject determines to what degree he/she has been facing the situation by selecting a percentage from 0% (never) to 100% (always), with 10% increments in between. Higher scores mean higher severity.
Time Frame: Baseline, 24 hours, 48 hrs, and 6 weeks (day 43)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | MIJ821 0.16 mg/kg Weekly | MIJ821 0.16 mg/kg Biweekly | MIJ821 0.32 mg/kg Weekly | MIJ821 0.32 mg/kg Biweekly | Ketamine 0.5 mg/kg Weekly | Placebo Weekly
Number analyzed (Participants) | 11 | 10 | 10 | 9 | 10 | 20
Scores on a Scale
  Adjusted arithmetic mean change from baseline at 24 hrs (n=11,10,10,9,10,20) | 1.82 (1.0) | 2.00 (1.1) | 1.20 (1.1) | 7.22 (1.1) | 2.10 (1.1) | 2.50 (0.8)
  Adjusted arithmetic mean change from baseline at 48 hrs (n=9,10,9,7,4,19): number analyzed (Participants) | 9 | 10 | 9 | 7 | 4 | 19
  Adjusted arithmetic mean change from baseline at 48 hrs (n=9,10,9,7,4,19) | 1.80 (1.1) | 2.30 (1.1) | 1.89 (1.1) | 3.46 (1.2) | 1.89 (1.4) | 2.43 (0.8)
  Adjusted arithmetic mean change from baseline at day 43 (n=8,8,8,6,9,17): number analyzed (Participants) | 8 | 8 | 8 | 6 | 9 | 17
  Adjusted arithmetic mean change from baseline at day 43 (n=8,8,8,6,9,17) | 1.38 (1.1) | 1.61 (1.1) | 1.02 (1.1) | 0.24 (1.3) | 1.86 (1.1) | 2.63 (0.8)

14. Secondary Outcome: Sheehan Suicidality Tracking Scale - (SSTS)
Description: Sheehan suicidality tracking scale(S-STS) is a fourteen-item (up to 22) scale. Each item in the S-STS is scored on a 5-point Likert scale (0=not at all, 1= a little, 2=moderately, 3=very, and 4=extremely). Data from the S-STS will be analyzed as individual item scores, suicidal ideation subscale score (sum of scores from items 2, 3 and 4, plus score from item 5 if ≤1), suicidal behavior subscale score (sum of scores from items 6, 7a and 8, plus score from item 5 if >1). Higher scores represent a more severe condition.
Time Frame: Change from baseline at 24 hours, 48 hours, and 6 weeks (Day 43)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | MIJ821 0.16 mg/kg Weekly | MIJ821 0.16 mg/kg Biweekly | MIJ821 0.32 mg/kg Weekly | MIJ821 0.32 mg/kg Biweekly | Ketamine 0.5 mg/kg Weekly | Placebo Weekly
Number analyzed (Participants) | 11 | 10 | 10 | 9 | 10 | 20
Scores on a Scale
  Suicidal behavior subscale score - Change at 24 hrs (n=11,10,10,9,10,20) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.11 (0.333) | -0.10 (0.316) | 0.00 (0.00)
  Suicidal behavior subscale score - Change at 48 hrs (n=9,10,9,7,4,19): number analyzed (Participants) | 9 | 10 | 9 | 7 | 4 | 19
  Suicidal behavior subscale score - Change at 48 hrs (n=9,10,9,7,4,19) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Suicidal behavior subscale score - Change at day 43 (n=8,8,8,6,9,17): number analyzed (Participants) | 8 | 8 | 8 | 6 | 9 | 17
  Suicidal behavior subscale score - Change at day 43 (n=8,8,8,6,9,17) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | -0.11 (0.333) | 0.12 (0.485)
  Suicidal ideation subscale score - Change at 24 hrs (n=11,10,10,9,10,20) | -0.45 (0.820) | -0.50 (0.850) | -0.30 (0.675) | 0.11 (1.269) | -0.40 (0.966) | -0.20 (0.523)
  Suicidal ideation subscale score - Change at 48 hrs (n=9,10,9,7,4,19): number analyzed (Participants) | 9 | 10 | 9 | 7 | 4 | 19
  Suicidal ideation subscale score - Change at 48 hrs (n=9,10,9,7,4,19) | -0.22 (0.667) | -0.50 (0.850) | -0.33 (0.707) | -0.43 (0.787) | 0.00 (0.00) | -0.16 (0.375)
  Suicidal ideation subscale score - Change at day 43 (n=8,8,8,6,9,17): number analyzed (Participants) | 8 | 8 | 8 | 6 | 9 | 17
  Suicidal ideation subscale score - Change at day 43 (n=8,8,8,6,9,17) | -0.38 (0.744) | -0.13 (0.354) | -0.13 (1.126) | 0.00 (1.265) | -0.11 (1.269) | 0.12 (1.111)
  SSTS total score - Change at 24 hrs (n=11,10,10,9,10,20) | -0.45 (0.820) | -0.50 (0.850) | -0.30 (0.675) | 0.11 (1.764) | -0.50 (1.269) | -0.20 (0.523)
  SSTS total score Change at 48 hrs (n=9,10,9,7,4,19): number analyzed (Participants) | 9 | 10 | 9 | 7 | 4 | 19
  SSTS total score Change at 48 hrs (n=9,10,9,7,4,19) | -0.22 (0.667) | -0.50 (0.850) | -0.33 (0.707) | -0.57 (1.134) | 0.00 (0.00) | -0.16 (0.375)
  SSTS total score - Change at Day 43 (n=8,8,8,6,9,17): number analyzed (Participants) | 8 | 8 | 8 | 6 | 9 | 17
  SSTS total score - Change at Day 43 (n=8,8,8,6,9,17) | -0.38 (0.744) | -0.13 (0.354) | -0.13 (1.126) | -0.17 (1.602) | -0.22 (1.563) | 0.47 (2.503)

15. Secondary Outcome: Percentage of Participants With Treatment Remissions (MADRS<7)
Description: Percentage of Participants with treatment remissions as assessed via (MADRS<7)
Time Frame: 24 hours, 48 hours, and 6 weeks (Day 43)
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | MIJ821 0.16 mg/kg Weekly | MIJ821 0.16 mg/kg Biweekly | MIJ821 0.32 mg/kg Weekly | MIJ821 0.32 mg/kg Biweekly | Ketamine 0.5 mg/kg Weekly | Placebo Weekly
Number analyzed (Participants) | 11 | 10 | 10 | 9 | 10 | 20
Percentage of Participants
  % of participants with remission at 24 hrs (n=11,10,10,8,10,20): number analyzed (Participants) | 11 | 10 | 10 | 8 | 10 | 20
  % of participants with remission at 24 hrs (n=11,10,10,8,10,20) | 9.1 | 20.0 | 0 | 11.1 | 20.0 | 5.0
  % of participants with remission at 48 hrs (n=9,10,9,7,4,19): number analyzed (Participants) | 9 | 10 | 9 | 7 | 4 | 19
  % of participants with remission at 48 hrs (n=9,10,9,7,4,19) | 22.2 | 10.0 | 11.1 | 28.6 | 25.0 | 10.5
  % of participants with remission at Day 43 (n=8,8,8,6, 9,17): number analyzed (Participants) | 8 | 8 | 8 | 6 | 9 | 17
  % of participants with remission at Day 43 (n=8,8,8,6, 9,17) | 25.0 | 37.5 | 0 | 16.7 | 22.2 | 11.8

16. Secondary Outcome: Change From Baseline in the Total Hamilton Anxiety Scale
Description: The Hamilton Anxiety Rating Scale (HAM-A) measures psychic anxiety and somatic anxiety symptoms based on a clinical assessment and patient interview. The scale has 14 items, with each item rated from 0-4, ranging from not present to very severe. A maximum score of 56 indicates the most severe case. (Hamilton 1959).
Time Frame: Baseline, and at 6 weeks (day 43)
Population: Intent-to-treat analysis set
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | MIJ821 0.16 mg/kg Weekly | MIJ821 0.16 mg/kg Biweekly | MIJ821 0.32 mg/kg Weekly | MIJ821 0.32 mg/kg Biweekly | Ketamine 0.5 mg/kg Weekly | Placebo Weekly
Number analyzed (Participants) | 8 | 8 | 8 | 6 | 8 | 17
Scores on a Scale | -1.94 (2.0) | -5.69 (2.0) | -7.17 (2.0) | -3.83 (2.2) | -4.93 (2.0) | -4.80 (1.4)

17. Secondary Outcome: Summary Statistics of Total Hamilton Anxiety Scale - Change From Baseline
Description: as for outcome 16
Time Frame: Change from baseline at week 6 (Day 43)
Population: Intent-to-treat analysis set
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | MIJ821 0.16 mg/kg Weekly | MIJ821 0.16 mg/kg Biweekly | MIJ821 0.32 mg/kg Weekly | MIJ821 0.32 mg/kg Biweekly | Ketamine 0.5 mg/kg Weekly | Placebo Weekly
Number analyzed (Participants) | 8 | 8 | 8 | 6 | 8 | 17
Scores on a Scale | -2.6 (6.927) | -5.4 (4.565) | -6.8 (6.606) | -4.2 (9.432) | -5.4 (7.763) | -5.1 (5.651)

18. Secondary Outcome: Change From Baseline in the Total Koukopoulos Mixed Depression Rating Scale
Description: The Koukopoulos Mixed Depression Rating Scale (KMDRS) assesses the excitatory or mixed nature in patients suffering from a Major Depressive Episode (MDE) as defined by DSM-5 criteria. This scale is meant to be used in conjunction with another scale that assess typical depression and anxiety symptoms. The scale contains 14 items to be evaluated by clinical assessment and patient interview on symptoms potentially experienced over the past week. Overall score increases with severity of symptoms and has a maximum score of 51. (Sani et al 2018).
Time Frame: Baseline, 24 hours, 48 hrs, and 6 weeks (day 43)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | MIJ821 0.16 mg/kg Weekly | MIJ821 0.16 mg/kg Biweekly | MIJ821 0.32 mg/kg Weekly | MIJ821 0.32 mg/kg Biweekly | Ketamine 0.5 mg/kg Weekly | Placebo Weekly
Number analyzed (Participants) | 11 | 10 | 10 | 9 | 10 | 20
Scores on a Scale
  Adjusted arithmetic mean change from baseline at 24 hrs (n=11,10,10,9,10,20) | -2.79 (0.9) | -2.38 (0.9) | -1.50 (1.0) | -2.46 (1.0) | -1.28 (1.0) | -2.33 (0.7)
  Adjusted arithmetic mean change from baseline at 48 hrs (n=9,10,9,7,4,19): number analyzed (Participants) | 9 | 10 | 9 | 7 | 4 | 19
  Adjusted arithmetic mean change from baseline at 48 hrs (n=9,10,9,7,4,19) | -2.95 (1.0) | -1.03 (0.9) | -1.97 (1.0) | -3.43 (1.1) | 0.01 (1.3) | -1.97 (0.7)
  Adjusted arithmetic mean change from baseline at day 43 (n=8,8,8,6,9,17): number analyzed (Participants) | 8 | 8 | 8 | 6 | 9 | 17
  Adjusted arithmetic mean change from baseline at day 43 (n=8,8,8,6,9,17) | -1.18 (1.0) | -1.06 (1.0) | -1.55 (1.1) | -2.04 (1.2) | -1.68 (1.0) | -1.59 (0.7)

19. Secondary Outcome: Responders (>50% Improvement in Bech-Rafaelsen Melancholia Scale) and Melancholia and Mixed Depression Checklist Factor.
Description: Percentage of Participants who responded. The first mixed depression checklist, created by Koukopoulos, has 8 criteria, which are marked as present or absent. If 3 or more criteria are marked present, then mixed depression would be diagnosed. The second mixed depression checklist, created by Angst, lists the 7 criteria for mania from DSM-5, which are marked as present or absent. If 3 or more criteria are marked present, excluding any duration criterion, then mixed depression would be diagnosed. The melancholia checklist, created by Ghaemi for this study, has 4 criteria, which are marked as present or absent. If 3 or more criteria are marked present, then melancholia would be diagnosed.
Time Frame: 24 hours, 48 hours, and 6 weeks (Day 43)
Population: Intent-to-treat analysis set. The sampling size for this outcome measure was too small to support inferential statistics; therefore, the results for this outcome measure were limited to this high-level summary table, where data for the 2 drugs were pooled (MIJ821, all doses and all dosage regimes) and Ketamine vs placebo.
Measure: Number; unit: Percentage of Participants
Groups:
- Koukopoulos: Koukopoulos Mixed Depression Rating Scale
- Angst: Mixed depression checklist, created by Angst
- Ghaemi: Melancholia checklist, created by Ghaemi
Arm/Group | Koukopoulos | Angst | Ghaemi
Number analyzed (Participants) | 9 | 9 | 9
Percentage of Participants
  % of participants who responded at 24 hrs - drugs (n=5,5,5): number analyzed (Participants) | 5 | 5 | 5
  % of participants who responded at 24 hrs - drugs (n=5,5,5) | 40.0 | 0 | 20.0
  % of participants who responded at 24 hrs - placebo (n=1,1,1): number analyzed (Participants) | 1 | 1 | 1
  % of participants who responded at 24 hrs - placebo (n=1,1,1) | 0 | 0 | 100
  % of participants who responded at 48 hrs - drugs (N=6, 6, 6): number analyzed (Participants) | 6 | 6 | 6
  % of participants who responded at 48 hrs - drugs (N=6, 6, 6) | 50.0 | 0 | 33.3
  % of participants who responded at 48 hrs - placebo (n=2,2,2): number analyzed (Participants) | 2 | 2 | 2
  % of participants who responded at 48 hrs - placebo (n=2,2,2) | 0 | 0 | 50.0
  % of participants who responded at Day 43 - drugs (n=9,9,9) | 55.6 | 0 | 44.4
  % of participants who responded at Day 43- placebo (n=3,3,3): number analyzed (Participants) | 3 | 3 | 3
  % of participants who responded at Day 43- placebo (n=3,3,3) | 33.3 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 30 post treatment, up to a maximum duration of 66 days.
Groups:
- MIJ821 0.16 mg/kg Weekly*: MIJ821 0.16 mg/kg weekly*
- MIJ821 0.16 mg/kg Every Other Week: MIJ821 0.16 mg/kg every other week
- MIJ821 0.32 mg/kg Every Other Week: MIJ821 0.32 mg/kg every other week
- Total: Total
Arm/Group | MIJ821 0.16 mg/kg Weekly* | MIJ821 0.16 mg/kg Every Other Week | MIJ821 0.32 mg/kg Weekly | MIJ821 0.32 mg/kg Every Other Week | Ketamine 0.5 mg/kg Weekly | Placebo Weekly | Total
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10 | 0/10 | 0/9 | 0/10 | 0/20 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/11 | 1/10 | 0/10 | 3/9 | 0/10 | 1/20 | 5/70
Other Adverse Events (participants affected / at risk) | 7/11 | 6/10 | 7/10 | 6/9 | 6/10 | 5/20 | 37/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MIJ821 0.16 mg/kg Weekly* (N=11) | MIJ821 0.16 mg/kg Every Other Week (N=10) | MIJ821 0.32 mg/kg Weekly (N=10) | MIJ821 0.32 mg/kg Every Other Week (N=9) | Ketamine 0.5 mg/kg Weekly (N=10) | Placebo Weekly (N=20) | Total (N=70)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Major depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Suicide threat (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MIJ821 0.16 mg/kg Weekly* (N=11) | MIJ821 0.16 mg/kg Every Other Week (N=10) | MIJ821 0.32 mg/kg Weekly (N=10) | MIJ821 0.32 mg/kg Every Other Week (N=9) | Ketamine 0.5 mg/kg Weekly (N=10) | Placebo Weekly (N=20) | Total (N=70)
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hyperacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2
Asthenopia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 2 | 0 | 4
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 2 | 1 | 1 | 1 | 5
Feeling abnormal (General disorders) | 3 | 1 | 2 | 0 | 0 | 0 | 6
Feeling of relaxation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Poisoning deliberate (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Blood potassium decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 2 | 1 | 0 | 0 | 0 | 0 | 3
Blood pressure systolic increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Akathisia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Amnesia (Nervous system disorders) | 2 | 0 | 5 | 3 | 0 | 0 | 10
Ataxia (Nervous system disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 3
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 3 | 1 | 1 | 2 | 1 | 10
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 2 | 1 | 1 | 1 | 6
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 2
Memory impairment (Nervous system disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 3
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 3
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Somnolence (Nervous system disorders) | 2 | 1 | 4 | 0 | 1 | 0 | 8
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Tunnel vision (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Abnormal dreams (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 3
Daydreaming (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Depersonalisation/derealisation disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 5 | 0 | 5
Disinhibition (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dissociation (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 3
Dissociative amnesia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Euphoric mood (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Illusion (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 3
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Mood swings (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Sleep terror (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Time perception altered (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/29/NCT03756129/Prot_001.pdf
  • Statistical Analysis Plan (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/29/NCT03756129/SAP_000.pdf